CLINICAL TRIAL: NCT06196905
Title: An Exploratory Study of MT-2990 in Patients With Antineutrophil Cytoplasmic Antibody (ANCA) -Associated Vasculitis (AAV)
Brief Title: An Exploratory Study of MT-2990 in Patients With AAV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT-2990-C-101; jRCT2031230538 (Other: Japan Registry of Clinical Trials (jRCT))
Record Dates: First submitted 2023-12-25; First posted 2024-01-09 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Antineutrophil Cytoplasmic Antibody (ANCA) -Associated Vasculitis (AAV)

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- MT-2990 (Experimental): MT-2990 will be administered intravenously every 4 weeks for a total of 6 doses.
  Interventions: Drug: MT-2990

INTERVENTIONS:
Drug: MT-2990 — i.v. infusion

SUMMARY:
To explore the efficacy, safety, pharmacokinetics and mechanism of action of MT-2990 in patients with AAV.

DETAILED DESCRIPTION:
Target sample size is 5~10 subjects administered MT-2990

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years or older on the day of informed consent
2. Clinical diagnosis of microscopic polyangiitis (MPA), granulomatosis with polyangiitis (GPA), or eosinophilic granulomatosis with polyangiitis (EGPA) according to 2022 ACR/EULAR Classification Criteria by the date of informed consent
3. Patients who meet at least one of the following criteria 1) or 2)

1) Patients is judged to be indicative of disease activity by the investigator with disease activity satisfying all of the following criteria at screening. If measurements or tests were performed multiple times during the screening period, the results from the latest date should be used to confirm that the criteria are met.

I. As elevated CRP due to active AAV, CRP >= 0.2 mg/dL

II. BVAS >= 1

III. At least one of the findings in a) to e) below. c) is only applicable to patients with EGPA.

1. FDG-PET/CT image finding(s) (Grade >= 2 [defined as FDG uptake = liver], and judged that the findings indicate inflammation by radiologist)
2. FVC(mL) below the lower limit of normal calculated using the "new reference range for Japanese using LMS method" and KL-6 >= 500 U/mL
3. History or presence of asthma and eosinophils counts >= 1000/µL
4. eGFR < 60 mL/min/1.73 m 2 and first-morning urine protein/creatinine ratio > 0.2 g/g Cr
5. Presence of hearing loss due to active AAV and air conduction hearing threshold (average of measurements at 0.25,0.5,1, 2, and 4 kHz) >= 30 dB in at least one ear

   2) Steroid-dependent patients who satisfy the following criteria I and II:

   I. Worsening of the primary disease due to steroid dose reduction or discontinuation within 6 months before the start of screening period, and then the steroid dose has been maintained at a level exceeding the time point of the worsening. Patients who meet only 2) of the inclusion criteria (3) must be judged by the investigator to be eligible to attempt to discontinue the steroid or reduce the steroid dose to the level at the worsening due to steroid dose reduction by Week 16 in principle.

   II. No initiation or increased dose of azathioprine or avacopan since the time of the worsening of the primary disease of I.

   Exclusion Criteria:
   1. Patients who have manifestations leading to life-threatening or vital organ dysfunction due to AAV, in the opinion of the Investigator.
   2. Patients with autoimmune diseases or vasculitis other than AAV such as systemic lupus erythematosus, IgA vasculitis, rheumatoid vasculitis, Sjogren's syndrome, anti-glomerular basement membrane nephritis, cryoglobulinemic vasculitis, idiopathic inflammatory muscle disease, systemic sclerosis.
   3. Patients who are judged by the Investigator to have an improvement trend of active finding(s) for AAV during remission maintenance treatment from the 12 weeks prior to the start of screening to the time of the first dose, and to be expected to improve spontaneously without change of treatment.
   4. Patients who received rituximab or immunosuppressive biologics (eg., TNF inhibitors) from 12 weeks prior to the start of screening to the time of the first dose.
   5. Patients who received mepolizumab from 8 weeks prior to the start of screening to the time of the first dose.
   6. Patients who received cyclophosphamide, methotrexate, mycophenolate mofetil, plasma exchange therapy or other immunosuppressive therapy from 4 weeks prior to screening to the time of the first dose.
   7. Patients who received a live vaccine from 4 weeks before the date of the first dose to the time of the first dose.
   8. Patients who have received steroids at prednisolone equivalent doses of more than 20 mg/day, initiated steroids, or increased the dose of steroids from 4 weeks prior to the start of screening to the time of the first dose.

      Exceptionally, only for rituximab treatment failures are allowed to initiate steroids or increase steroids dose up to that of their most recent induction remission therapy (i.e., doses exceeding 20 mg/day of prednisolone equivalent are allowed) until the day before the first dose.
   9. Patients who have initiated, increased, or decreased the dose of azathioprine from 4 weeks prior to the start of screening to the time of the first dose.
   10. Patients who have initiated, increased, or decreased the dose of avacopan from 4 weeks prior to the start of screening to the time of the first dose.
   11. Patients with concomitant or history of hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV) infection unless patients have negative test result of hepatitis B virus surface (HBs) antigen, HBs antibody, and hepatitis B virus core (HBc) antibody at screening, or have maintained a negative HCV-RNA test result for at least 12 weeks after completion of hepatitis C treatment.
   12. Patients with systemic active infections at the day of screening evaluation or the date of the first dose.
   13. Patients with a history of malignancy within 5 years prior to the start of screening, except for basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or intraepithelial carcinoma of the cervix who have completed treatment (including therapy other than anticancer agents for the treatment of cancer) without recurrence for at least 1 year.
   14. History of anaphylaxis or clinically significant allergic symptoms due to administration of antibody products.
   15. Patients who have received anti-IL-33 antibodies including this investigational drug in the past.
   16. Patients with serious complications.
   17. Male and female patients of childbearing potential (Excluding postmenopausal women who have been amenorrheic for at least 1 year and women who have undergone surgical hysterectomy or bilateral oophorectomy) who are unable to obtain consent to use contraception from the date of consent until 12 weeks after completion of study drug administration.
   18. Female patients who are pregnant, breastfeeding, or possibly pregnant
   19. Patients who participated in any clinical trial and received the investigational medical product within 12 weeks (or 5 half-lives of investigational medical product, whichever is longer) prior to obtaining consent.
   20. Patients who are judged by the Investigator to be ineligible for this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2024-06-24 (Actual); Primary Completion 2026-01-14 (Actual); Study Completion 2026-01-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Birmingham Vasculitis Activity Score (BVAS) at each scheduled timepoints | Up to Week 24
  No primary endpoint is used, because various exploratory analyses are performed.
  Birmingham Vasculitis Activity Score (BVAS) form is divided into 9 organ-based systems, with each section including symptoms/signs that are typical of that particular organ involvement in systemic vasculitis. The clinician only scores features believed to be due to active vasculitis. Completion of the form provides a numerical score, which ranges from 0 (best health) to 63 (worst health).
Proportion of subjects who achieve BVAS=0 at each scheduled timepoints | Up to week 24
  No primary endpoint is used, because various exploratory analyses are performed.
Change from baseline in Vasculitis Damage Index (VDI) at each scheduled timepoints. | Up to week 24
  No primary endpoint is used, because various exploratory analyses are performed.
  Vasculitis Damage Index (VDI) is comprised of 64 items of damage, grouped into 11 organ-based systems or categorizations. Damage is defined as the presence of non-healing scars and does not give any indication of current disease activity. Damage is also defined as having been present or currently present for at least 3 months. Completion of the form provides a numerical score, which ranges from 0 (best health) to 64 (worst health).
Patient Global Impression of Change (PGIC) at each scheduled timepoints | Up to week 24
  No primary endpoint is used, because various exploratory analyses are performed.
  Patient Global Impression of Change (PGIC) is a questionnaire to evaluate the overall impression of improvement by patient from 1 (very much improved) to 7 (very much worse). Higher PGIC scores indicated worse outcome.
Clinical Global Impression of Change (CGIC) at each scheduled timepoints | Up to week 24
  No primary endpoint is used, because various exploratory analyses are performed.
  Clinician Global Impression of Change (CGIC) a questionnaire to evaluate the overall impression of improvement by clinician from 1 (very much improved) to 7 (very much worse). Higher CGIC scores indicated worse outcome.
Change from baseline in FDG-PET/CT findings at week 24 | Baseline and week 24
  No primary endpoint is used, because various exploratory analyses are performed.
Change from baseline in chest CT findings at each scheduled timepoints | Up to week 24
  No primary endpoint is used, because various exploratory analyses are performed.
Change from baseline in head and neck CT/MRI findings at each scheduled timepoints | Up to week 24
  No primary endpoint is used, because various exploratory analyses are performed.
Change from baseline in respiratory function tests (FVC [mL]) at each scheduled timepoints | Up to week 24
  No primary endpoint is used, because various exploratory analyses are performed.
Change from baseline in hearing threshold measured by pure-tone audiometry at each scheduled timepoints | Up to week 24
  No primary endpoint is used, because various exploratory analyses are performed.
Time course of BM {eGFR, urine protein/creatinine ratio (first morning urine), eosinophil count, serum KL-6, CRP, and ANCA-titer (MPO-ANCA, PR3-ANCA)} at each scheduled timepoints | Up to week 24
  No primary endpoint is used, because various exploratory analyses are performed.
Change in dosage of steroid | Up to week 24
  No primary endpoint is used, because various exploratory analyses are performed.
Change from baseline in SF-36 at each scheduled timepoints | Up to week 24
  No primary endpoint is used, because various exploratory analyses are performed.
Change from baseline in EQ-5D-5L at each scheduled timepoints | Up to week 24
  No primary endpoint is used, because various exploratory analyses are performed.

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Tanabe Pharma Corporation
Locations (8):
- Japan (8):
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Kagawa University Hospital, Kita-gun, Kagawa-ken
  - Saitama Medical University Hospital, Iruma-gun, Saitama
  - Saitama Medical Center, Kawagoe, Saitama
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - NHO Tokyo Medical Center, Meguro-ku, Tokyo
  - Kyorin University Hospital, Mitaka-shi, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo

IPD SHARING:
Plan to Share IPD: No